CLINICAL TRIAL: NCT00007852
Title: A Phase II Trial of Rituxan and BEAM High-Dose Chemotherapy and Autologous Peripheral Blood Progenitor Transplant for Lymphoma
Brief Title: Rituximab & Combination Chemotherapy Followed by Transplantation in Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0045-00-FB; P30CA036727 (NIH); NCI-V00-1634 (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2001-01-06; First posted 2004-02-12 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Carmustine; Cytarabine; Etoposide; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): Rituxan and BEAM with autologous stem cell transplant
  Interventions: Biological: rituximab; Drug: carmustine; Drug: cytarabine; Drug: etoposide; Drug: melphalan; Procedure: autologous hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: rituximab — Rituximab at 375 mg/m2 administered approximately one week apart prior to collection of the hematopoietic stem cells. Rituxan at a dose of 375 mg/m2 IV will be given either on the days prior to initiation of the BCNU (days -10 to -7) or on the same day that the BCNU is administered for the BEAM chemotherapy regimen (Day -6). A fourth infusion of Rituxan 375 mg/m2 will be given at 30 day (+/- 20 days) post-transplant. At approximately 6 months post-transplant, if the patients have not had progressive lymphoma, they will receive four weekly doses of Rituxan 375 mg/m2 IV.
  Other Names: Rituxan
Drug: carmustine — BCNU 300 mg/M2 IV day -6
  Other Names: BCNU
Drug: cytarabine — 100 mg/m2 on days -5 through -2
  Other Names: BEAM chemotherapy regimen
Drug: etoposide — 100mg/M2 BID on days -5 through -2
  Other Names: BEAM chemotherapy regimen
Drug: melphalan — 140 mg/m2 IV on day -1
  Other Names: BEAM chemotherapy regimen
Procedure: autologous hematopoietic stem cell transplantation — Following the chemotherapy, on day 0 of treatment, the previously stored hematopoietic stem cells will be reinfused via the central venous line

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation or bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of rituximab and combination chemotherapy followed by bone marrow or peripheral stem cell transplantation in treating patients who have relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the complete and partial response rate of patients with relapsed or refractory B-cell non-Hodgkin's lymphoma treated with rituximab and high-dose carmustine, etoposide, cytarabine and melphalan followed by autologous bone marrow or peripheral blood stem cell transplantation. II. Determine the toxicity profile of this regimen in these patients. III. Compare the levels of soluble CD20 antigen and rituximab blood levels with patient outcomes in this patient population.

OUTLINE: Patients receive two doses of rituximab IV over 3-4 hours 1 week apart. Stem cells from the peripheral blood or bone marrow are collected at least 1 week after the second dose of rituximab. Following stem cell collection, patients receive a third dose of rituximab IV as above between days -10 and -6. Patients then receive high-dose chemotherapy consisting of carmustine IV on day -6, etoposide IV twice daily and cytarabine IV on days -5 to -2, and melphalan IV on day -1. On day 0 patients undergo autologous bone marrow or peripheral blood stem cell transplantation. After transplantation, patients receive a fourth dose of rituximab as above at approximately day 30, and then weekly over 4 weeks at approximately 6 months in the absence of disease progression or unacceptable toxicity. Patients are followed at 1 year and then annually thereafter.

PROJECTED ACCRUAL: A total of 23-40 patients will be accrued for this study within 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CD20-positive B-cell non-Hodgkin's lymphoma
* Transplantation candidate
* Primary induction failure
* Chemotherapy refractory disease
* Received at least 3 prior chemotherapy regimens or diagnosis of mantle cell lymphoma
* Age 19 and over
* Performance status: WHO 0-2
* Life expectancy at least 6 months
* Absolute neutrophil count at least 1,000/mm3 (unless due to lymphomatous involvement of the marrow)
* Platelet count more than 50,000/mm3 (unless due to lymphomatous involvement of the marrow)
* Hemoglobin more than 9.0 g/dL (unless due to lymphomatous involvement of the marrow)
* Fertile patients must use effective contraception
* Concurrent non-steroidal hormones for non-lymphoma-related conditions (e.g., insulin for diabetes) allowed

Exclusion Criteria:

* No other concurrent chemotherapy
* No concurrent corticosteroids except for transient control or prevention of nausea or vomiting
* No concurrent external beam radiotherapy during transplantation therapy
* No other concurrent antitumoral or investigational agents
* No history of T-cell lymphoma
* No relapse or progression after rituximab therapy within 3 months before transplantation
* No serious disease or condition that would preclude study
* Not pregnant or nursing/negative pregnancy test

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2000-09-01 (Actual); Primary Completion 2002-01-01 (Actual); Study Completion 2011-01-01 (Actual)

PRIMARY OUTCOMES:
100 day (complete + partial) response rate | 100 days
  The primary endpoint for this study is 100 day (complete + partial) response rate

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Vose, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States